CLINICAL TRIAL: NCT04333004
Title: Analysis of Gut Microbiota in Patients With Brain Metastasis of Non-small Cell Lung Cancer Treated by Pembrolizumab Combined With Chemotherapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiaorong Dong (Other)
Responsible Party: Sponsor-Investigator, Xiaorong Dong, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Gut Microbiota; NSCLC; Pembrolizumab; Chemotherapy
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab Combined With Chemotherapy (Experimental)
  Interventions: Drug: Pembrolizumab Combined With Chemotherapy

INTERVENTIONS:
Drug: Pembrolizumab Combined With Chemotherapy — Pembrolizumab and chemotherapy are carried out at the same time for every 3 weeks

SUMMARY:
Analysis of Gut Microbiota in Patients With Brain Metastasis of Non-small Cell Lung Cancer Treated by Pembrolizumab Combined With Chemotherapy

ELIGIBILITY:
Inclusion Criteria:

- non-small cell lung cancer patients with less than brain metastases Patients must have received at least the first-line anti-tumor treatment, and the front-line treatment must include chemotherapy or targeted treatment with a platinum containing combination scheme, but not anti-PD-1 / L1 treatment Patients who have not received intracranial local treatment before

Exclusion Criteria:

- Patients who toke major surgery within 4 weeks prior to enrollment or had ununited wounds Patients with hemorrhage in intracranial metastasis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
diversity of gut microbiota | 1 year
  Species and abundance of gut microbiota